CLINICAL TRIAL: NCT04665310
Title: Evaluation of Early Dose Escalation Using Extended-Release Tacrolimus (Envarsus XR®) to Reduce Acute Rejection and Donor Specific Antibodies in African American Renal Transplant Recipients
Brief Title: Evaluation of Anti-rejection Drug, Tacrolimus, in African-Americans With Kidney Transplant
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Veloxis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Ahmed Osama Gaber, MD, Director, Houston Methodist J.C. Walter Jr. Transplant Center, The Methodist Hospital Research Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00018836
Record Dates: First submitted 2019-04-02; First posted 2020-12-11 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Kidney Disease, End-Stage; Donor Specific Antibodies; Acute Rejection of Renal Transplant
Keywords: Renal Transplant; Donor Specific Antibodies; African American; Acute Rejection of Renal Transplant; Kidney Transplant; End Stage Renal Disease
MeSH Terms: conditions — Kidney Failure, Chronic | interventions — Tacrolimus

STUDY DESIGN:
Intervention Model Description: Parallel Group - Dose Escalation with 2 groups stratified by pPRA <75% and >75% and then randomized into 3 Intensity Arms (Low, Moderate and High) based on dosing of Envarsus XR.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Group 1 - Low-Intensity (Active Comparator): All patients will receive standard induction immunosuppression according to institution protocol. TAC will be started when clinically appropriate according to institution protocol.
  TAC dosing will be 2 mg twice daily to be reduced by 20% after week 1 and start Envarsus XR once daily.
  Target Tacrolimus Trough Concentrations:
  Week 0 to Week 4: 8-10 mg/mL Month 1 to Month 3: 6-8 mg/mL
  Interventions: Drug: Envarsus XR
- Group 1 - Moderate-Intensity (Active Comparator): All patients will receive standard induction immunosuppression according to institution protocol. TAC will be started when clinically appropriate according to institution protocol.
  TAC dosing will be 3 mg twice daily to be reduced by 20% after week 1 and start Envarsus XR once daily.
  Target Tacrolimus Trough Concentrations:
  Week 0 to Week 4: 10-12 mg/mL Month 1 to Month 3: 8-10 mg/mL
  Interventions: Drug: Envarsus XR
- Group 1 - High-Intensity (Active Comparator): All patients will receive standard induction immunosuppression according to institution protocol. TAC will be started when clinically appropriate according to institution protocol.
  TAC dosing will be 4 mg twice daily to be reduced by 20% after week 1 and start Envarsus XR once daily.
  Target Tacrolimus Trough Concentrations:
  Week 0 to Week 4: 12-14 mg/mL Month 1 to Month 3: 10-12 mg/mL
  Interventions: Drug: Envarsus XR
- Group 2 - Low-Intensity (Active Comparator): All patients will receive standard induction immunosuppression according to institution protocol. TAC will be started when clinically appropriate according to institution protocol.
  TAC dosing will be 2 mg twice daily to be reduced by 20% after week 1 and start Envarsus XR once daily.
  Target Tacrolimus Trough Concentrations:
  Week 0 to Week 4: 8-10 mg/mL Month 1 to Month 3: 6-8 mg/mL
  Interventions: Drug: Envarsus XR
- Group 2 - Moderate-Intensity (Active Comparator): All patients will receive standard induction immunosuppression according to institution protocol. TAC will be started when clinically appropriate according to institution protocol.
  TAC dosing will be 3 mg twice daily to be reduced by 20% after week 1 and start Envarsus XR once daily.
  Target Tacrolimus Trough Concentrations:
  Week 0 to Week 4: 10-12 mg/mL Month 1 to Month 3: 8-10 mg/mL
  Interventions: Drug: Envarsus XR
- Group 2 - High-Intensity (Active Comparator): All patients will receive standard induction immunosuppression according to institution protocol. TAC will be started when clinically appropriate according to institution protocol.
  TAC dosing will be 4 mg twice daily to be reduced by 20% after week 1 and start Envarsus XR once daily.
  Target Tacrolimus Trough Concentrations:
  Week 0 to Week 4: 12-14 mg/mL Month 1 to Month 3: 10-12 mg/mL
  Interventions: Drug: Envarsus XR

INTERVENTIONS:
Drug: Envarsus XR — tacrolimus, extended-release tablets, a calcineurin inhibitor
  Other Names: Life Cycle Pharma (LCP)-tacrolimus; once-daily extended-release tacrolimus; once-daily prolonged-release tacrolimus; Tacrolimus-LCP

SUMMARY:
In spite of conventional immunosuppression with lymphocyte-depleting induction followed by tacrolimus- and mycophenolate-based regimens, African American (AA) renal transplant recipients experience higher rates of acute rejection (AR), donor specific antibodies (DSA), and graft failure. Envarsus Extended-Release (XR)® (ENV) is a novel extended-release formulation of tacrolimus with a favorable pharmacokinetic profile, even in the setting of CYP3A5*1 allele (rapid metabolizers). The investigator will evaluate the safety and efficacy of early dose escalation with ENV in AA recipients. The study hypothesis is that higher tacrolimus target concentrations may be achieved without typical dose-limiting toxicities, and this may ultimately result in lower incidence of early AR, DSA, and graft loss.

DETAILED DESCRIPTION:
Phase 4 (post-marketing) De novo African American living or deceased donor renal transplant recipients 18 to 65 years of age Number of subjects to be enrolled: 60

All patients will receive standard induction immunosuppression according to institution protocol. Within one week of transplantation, all patients will be converted from immediate-release tacrolimus (TAC) to extended-release tacrolimus (ENV) at 20% reduction in total daily dosage. Patients will be randomized to low-, moderate-, or high-intensity ENV groups, stratified by peak panel reactive antibody (pPRA) greater than or equal to 75%. Target tacrolimus trough concentrations for the first month post-transplant will be 8-10 ng/mL in low-intensity group, 10-12 ng/mL in moderate-intensity group, and 12-14 ng/mL in high-intensity group; likewise from month 1-3 post-transplant, target trough concentrations will be 6-8 ng/mL, 8-10 ng/mL, and 10-12 ng/mL, respectively. Subjects experiencing dose-limiting adverse events (AEs) will be de-escalated as warranted. Following month 3, all patients will be maintained on ENV at target tacrolimus trough concentrations according to institution protocol. Additional maintenance immunosuppression will consist of mycophenolate mofetil (MMF) at a goal dose of 2000 mg daily along with an oral prednisone taper to 5-10 mg daily by the end of month 1. All patients will be followed for 6 months post-transplant.

ELIGIBILITY:
Inclusion Criteria:

* • Primary live donor or deceased donor renal allograft

  * African American patients aged 18 to 65 years
  * Ability to take oral medications
  * Not currently on medications known to significantly interfere with tacrolimus metabolism, e.g. strong CYP3A4 inducers or inhibitors including but not limited to rifampin, rifabutin, phenytoin, carbamazepine, phenobarbital, protease inhibitors, azole antifungal (voriconazole, itraconazole, posaconazole, ketoconazole)

    o Note: All patients will be discharged on clotrimazole 10 mg three times daily for one month for thrush prophylaxis, a known mild-to-moderate CYP3A4 inhibitor
  * Female subjects of childbearing potential:

    * Not current pregnant
    * Agree not to try to become pregnant during the study period
    * Agree to consistently use two forms of highly effective birth control throughout the study period
  * Provision of signed and dated informed consent form
  * Stated willingness to comply with all study procedures and availability for the duration of the study

Exclusion Criteria:

* • Presence of a positive T- or B-cell flow cytometry allogeneic crossmatch

  * Presence of pre-formed anti-human leukocyte antigen (HLA) donor-specific antibodies (DSAs)
  * Recipient of an ABO-incompatible organ
  * Receipt of a multi-organ or dual kidney transplant
  * Receipt of pediatric en bloc deceased donor kidneys
  * Receipt of deceased donor kidney with a kidney donor profile index (KDPI) greater than or equal to 85%
  * Has undergone desensitization, or received antibody removal, anti-B-cell, or anti-plasma cell therapy in the 90 days preceding the transplant
  * Planned initiation of antibody removal (i.e. plasmapheresis) within 7 days of the transplant procedure
  * Positive test for latent tuberculosis (TB) and has not previously received adequate anti-microbial therapy or would require TB prophylaxis after transplant
  * Uncontrolled concomitant infection that would not allow for targeting escalated tacrolimus trough concentrations, as deemed by prescriber
  * Known infection or seropositivity for hepatitis B virus (HBV, defined by positive HBsAg, anti-HBcAg, or positive viral load) or hepatitis C virus (HCV) with active viral load
  * Current malignancy
  * Use of an investigational study in the 30 days prior to the transplant procedure

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2018-09-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants reaching the composite endpoint | 6 months
  Composite endpoint of freedom from all of the following: i) biopsy-proven T-cell mediated rejection Banff Grade ≥1A, ii) antibody-mediated rejection, iii) de novo DSA, or iv) immune-mediated graft loss. The endpoint is a binary endpoint (Yes or No) of the composite of all 4 potential outcomes. The presence of any one of the four possible outcomes will be counted as a No for the binary endpoint (no freedom from the composite endpoint). The absence of all 4 possible outcomes will be counted as Yes for freedom from all of the possible outcomes.

SECONDARY OUTCOMES:
Proportion of subjects experiencing nephrotoxicity during the study | 6 months
  Increase in serum creatinine of ≥0.3mg/dL
Proportion of subjects experiencing neurotoxicity during the study | 6 months
  Clinical intolerability including headache or significant tremors that resolve with reduction of the dose of Envarsus
Proportion of subjects experiencing infectious complications during the study | 6 months
  Participants requiring extended (>2 weeks) reduction in dose of Envarsus due to BK-polyomavirus or cytomegalovirus viral loads at 1, 3, and 6 months post-transplant
Difference in estimated glomerular filtration rate at 1, 3, and 6 months between groups of enrolled subjects | 6 months
  Assessed as the Chronic Kidney Disease - Epidemiology Collaboration equation
Difference in immunosuppressant side effects between enrolled subjects | 6 months
  Assessed using the "Immunosuppressant Side Effects Instrument - The Memphis Survey" questionnaire
Enrolled subject overall survival and Graft survival at 6 months | 6 months
  Freedom from death and from graft loss at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed O Gaber, MD, Principal Investigator — Houston Methodist Physicians Organization

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kidney Disease: Improving Global Outcomes (KDIGO) Transplant Work Group. KDIGO clinical practice guideline for the care of kidney transplant recipients. Am J Transplant. 2009 Nov;9 Suppl 3:S1-155. doi: 10.1111/j.1600-6143.2009.02834.x. PMID 19845597
- [Background] Young CJ, Gaston RS. Renal transplantation in black Americans. N Engl J Med. 2000 Nov 23;343(21):1545-52. doi: 10.1056/NEJM200011233432107. No abstract available. PMID 11087885
- [Background] Narayanan M, Pankewycz O, Shihab F, Wiland A, McCague K, Chan L. Long-term outcomes in African American kidney transplant recipients under contemporary immunosuppression: a four-yr analysis of the Mycophenolic acid Observational REnal transplant (MORE) study. Clin Transplant. 2014 Feb;28(2):184-91. doi: 10.1111/ctr.12294. Epub 2013 Dec 24. PMID 24372743
- [Background] Lamb KE, Lodhi S, Meier-Kriesche HU. Long-term renal allograft survival in the United States: a critical reappraisal. Am J Transplant. 2011 Mar;11(3):450-62. doi: 10.1111/j.1600-6143.2010.03283.x. Epub 2010 Oct 25. PMID 20973913
- [Background] Patel SJ, Suki WN, Loucks-DeVos J, Graviss EA, Nguyen DT, Knight RJ, Kuten SA, Moore LW, Teeter LD, Gaber LW, Gaber AO. Disparate rates of acute rejection and donor-specific antibodies among high-immunologic risk renal transplant subgroups receiving antithymocyte globulin induction. Transpl Int. 2016 Aug;29(8):897-908. doi: 10.1111/tri.12791. Epub 2016 Jul 7. PMID 27196395
- [Background] Bunnapradist S, Ciechanowski K, West-Thielke P, Mulgaonkar S, Rostaing L, Vasudev B, Budde K; MELT investigators. Conversion from twice-daily tacrolimus to once-daily extended release tacrolimus (LCPT): the phase III randomized MELT trial. Am J Transplant. 2013 Mar;13(3):760-9. doi: 10.1111/ajt.12035. Epub 2012 Dec 21. PMID 23279614
- [Background] Budde K, Bunnapradist S, Grinyo JM, Ciechanowski K, Denny JE, Silva HT, Rostaing L; Envarsus study group. Novel once-daily extended-release tacrolimus (LCPT) versus twice-daily tacrolimus in de novo kidney transplants: one-year results of Phase III, double-blind, randomized trial. Am J Transplant. 2014 Dec;14(12):2796-806. doi: 10.1111/ajt.12955. Epub 2014 Oct 2. PMID 25278376
- [Background] Gaber AO, Alloway RR, Bodziak K, Kaplan B, Bunnapradist S. Conversion from twice-daily tacrolimus capsules to once-daily extended-release tacrolimus (LCPT): a phase 2 trial of stable renal transplant recipients. Transplantation. 2013 Jul 27;96(2):191-7. doi: 10.1097/TP.0b013e3182962cc1. PMID 23715050
- [Background] Bunnapradist S, Rostaing L, Alloway RR, West-Thielke P, Denny J, Mulgaonkar S, Budde K. LCPT once-daily extended-release tacrolimus tablets versus twice-daily capsules: a pooled analysis of two phase 3 trials in important de novo and stable kidney transplant recipient subgroups. Transpl Int. 2016 May;29(5):603-11. doi: 10.1111/tri.12770. Epub 2016 Apr 3. PMID 26953629
- [Background] Trofe-Clark J, Brennan DC, West-Thielke P, Milone MC, Lim MA, Neubauer R, Nigro V, Bloom RD. Results of ASERTAA, a Randomized Prospective Crossover Pharmacogenetic Study of Immediate-Release Versus Extended-Release Tacrolimus in African American Kidney Transplant Recipients. Am J Kidney Dis. 2018 Mar;71(3):315-326. doi: 10.1053/j.ajkd.2017.07.018. Epub 2017 Nov 20. PMID 29162334
- [Background] Langone A, Steinberg SM, Gedaly R, Chan LK, Shah T, Sethi KD, Nigro V, Morgan JC; STRATO Investigators. Switching STudy of Kidney TRansplant PAtients with Tremor to LCP-TacrO (STRATO): an open-label, multicenter, prospective phase 3b study. Clin Transplant. 2015 Sep;29(9):796-805. doi: 10.1111/ctr.12581. Epub 2015 Aug 6. PMID 26113208
- [Background] Kuypers DR, Claes K, Evenepoel P, Maes B, Vanrenterghem Y. Clinical efficacy and toxicity profile of tacrolimus and mycophenolic acid in relation to combined long-term pharmacokinetics in de novo renal allograft recipients. Clin Pharmacol Ther. 2004 May;75(5):434-47. doi: 10.1016/j.clpt.2003.12.009. PMID 15116056
- [Background] Winsett RP, Arheart K, Stratta RJ, Alloway R, Wicks MN, Gaber AO, Hathaway DK. Evaluation of an immunosuppressant side effect instrument. Prog Transplant. 2004 Sep;14(3):210-6, 240. doi: 10.1177/152692480401400306. PMID 15495780
- [Background] Staatz CE, Tett SE. Clinical pharmacokinetics and pharmacodynamics of tacrolimus in solid organ transplantation. Clin Pharmacokinet. 2004;43(10):623-53. doi: 10.2165/00003088-200443100-00001. PMID 15244495
- [Background] Kuypers DR, Peeters PC, Sennesael JJ, Kianda MN, Vrijens B, Kristanto P, Dobbels F, Vanrenterghem Y, Kanaan N; ADMIRAD Study Team. Improved adherence to tacrolimus once-daily formulation in renal recipients: a randomized controlled trial using electronic monitoring. Transplantation. 2013 Jan 27;95(2):333-40. doi: 10.1097/TP.0b013e3182725532. PMID 23263559
- [Background] Ho ET, Wong G, Craig JC, Chapman JR. Once-daily extended-release versus twice-daily standard-release tacrolimus in kidney transplant recipients: a systematic review. Transplantation. 2013 May 15;95(9):1120-8. doi: 10.1097/TP.0b013e318284c15b. PMID 23542469
- [Background] Beckebaum S, Iacob S, Sweid D, Sotiropoulos GC, Saner F, Kaiser G, Radtke A, Klein CG, Erim Y, de Geest S, Paul A, Gerken G, Cicinnati VR. Efficacy, safety, and immunosuppressant adherence in stable liver transplant patients converted from a twice-daily tacrolimus-based regimen to once-daily tacrolimus extended-release formulation. Transpl Int. 2011 Jul;24(7):666-75. doi: 10.1111/j.1432-2277.2011.01254.x. Epub 2011 Apr 5. PMID 21466596
- [Background] Doesch AO, Mueller S, Konstandin M, Celik S, Erbel C, Kristen A, Frankenstein L, Koch A, Dengler TJ, Ehlermann P, Zugck C, De Geest S, Katus HA. Increased adherence after switch from twice daily calcineurin inhibitor based treatment to once daily modified released tacrolimus in heart transplantation: a pre-experimental study. Transplant Proc. 2010 Dec;42(10):4238-42. doi: 10.1016/j.transproceed.2010.09.074. PMID 21168673
- [Background] Maldonado G, Greenland S. Simulation study of confounder-selection strategies. Am J Epidemiol. 1993 Dec 1;138(11):923-36. doi: 10.1093/oxfordjournals.aje.a116813. PMID 8256780
- [Background] Wasserman L. Bayesian Model Selection and Model Averaging. J Math Psychol. 2000 Mar;44(1):92-107. doi: 10.1006/jmps.1999.1278. PMID 10733859